CLINICAL TRIAL: NCT02611986
Title: Evaluation of Video Laryngoscopy (Video Macintosh-blade) and Direct Laryngoscopy (EMMA-Study): A Prospective, Randomized Trial
Brief Title: Evaluation of Video Laryngoscopy (Video Macintosh-blade) and Direct Laryngoscopy (EMMA-Study)
Acronym: EMMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Collaborators: Western University, Canada (Other); Mutterhaus der Borromäerinnen, Germany (Unknown); Christophorus Hospital, Germany (Unknown)
Responsible Party: Principal Investigator, Marc Kriege, MD, MD, Johannes Gutenberg University Mainz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JohannesGUE
Record Dates: First submitted 2015-11-15; First posted 2015-11-23 (Estimated); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Airway Morbidity
Keywords: Airway management; video laryngoscope

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- McGrath MAC (Experimental): tracheal intubation using the McGrath MAC
  Interventions: Device: the McGrath MAC
- Macintosh Laryngoscope (Experimental): tracheal intubation using the Macintosh Laryngoscope
  Interventions: Device: the Macintosh Laryngoscope

INTERVENTIONS:
Device: the McGrath MAC — in a randomised order we evaluate the success rate with the first attempt of the tracheal tube into the trachea.
  Arms: McGrath MAC
Device: the Macintosh Laryngoscope — in a randomised order we evaluate the success rate with the first attempt of the tracheal tube into the trachea.
  Arms: Macintosh Laryngoscope

SUMMARY:
A randomized controlled prospective study of laryngoscopy and intubation success comparing direct laryngoscopy and the McGrath® Mac videolaryngoscope.

DETAILED DESCRIPTION:
As airway management continues to evolve the investigators do not have an accurate statement of the success of direct laryngoscopy in daily clinical practice. The use of videolaryngoscopy is increasing as a technique for rescue intubation as well as for elective intubation. Current airway management guidelines recommend video-assisted laryngoscopy as a choice for basic airway management. This is a proposed comparison study of a video laryngoscope, use in the daily anesthesia practice, and its likely increased success compared to direct laryngoscopy. An international, multi-center, prospective randomized comparative trial (RCT) is proposed testing the superiority of oral tracheal intubation with the McGrath® MAC versus conventional laryngoscope in adult patients under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 Years No concurrent participation in another study
* capacity to consent
* Present written informed consent of the research participant
* Elective surgery under general anesthesia

Exclusion Criteria:

* Age <18 years
* Existing pregnancy
* Lack of consent
* inability to consent
* emergency patients
* Emergency situations in the context of a Difficult Airway Management
* ASA classification> 3
* situations where the possibility of accumulated gastric contents
* Participation in another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2466 (Actual)
Dates: Start 2015-11-11 (Actual); Primary Completion 2019-05-07 (Actual); Study Completion 2019-05-14 (Actual)

PRIMARY OUTCOMES:
intubation success | at intubation; < 120 seconds
  successful tracheal intubation at the first attempt, compared to more than one attempt

SECONDARY OUTCOMES:
Cormack and Lehane Classification | < 120 seconds
  after insert the instrument the user describe the view of the laryngeal structure
Percentage of glottic opening | < 120 seconds
  airway visualization during intubation process
Number of attempts | < 120 seconds
  after two attempts using defined rescue techniques (e.g. rigid stylet, laryngeal mask)
IDS (intubation difficult score) | < 120 seconds
  intubation difficult score

CONTACTS AND LOCATIONS:
Overall Officials: Marc Kriege, MD, Principal Investigator — University JG, Mainz; Rüdiger Noppens, MD,Phd, Principal Investigator — Western University
Locations (1):
- Department of Anesthesiology,Prof. C. Werner, Universitätsmedizin of the JG University, Mainz, Rhineland-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wallace CD, Foulds LT, McLeod GA, Younger RA, McGuire BE. A comparison of the ease of tracheal intubation using a McGrath MAC((R)) laryngoscope and a standard Macintosh laryngoscope. Anaesthesia. 2015 Nov;70(11):1281-5. doi: 10.1111/anae.13209. Epub 2015 Sep 4. PMID 26336853
- [Background] Alvis BD, Hester D, Watson D, Higgins M, St Jacques P. Randomized controlled trial comparing the McGrath MAC video laryngoscope with the King Vision video laryngoscope in adult patients. Minerva Anestesiol. 2016 Jan;82(1):30-5. Epub 2015 Apr 17. PMID 25881731
- [Derived] Kriege M, Alflen C, Tzanova I, Schmidtmann I, Piepho T, Noppens RR. Evaluation of the McGrath MAC and Macintosh laryngoscope for tracheal intubation in 2000 patients undergoing general anaesthesia: the randomised multicentre EMMA trial study protocol. BMJ Open. 2017 Aug 21;7(8):e016907. doi: 10.1136/bmjopen-2017-016907. PMID 28827261